CLINICAL TRIAL: NCT03220139
Title: Type of Dietary Fat Intakes in Relation to Mortality in US Adults: An Iso-caloric Substitution Analysis From the American National Health and Nutrition Examination Survey Linked to the US Mortality Registry
Status: Completed | Type: Observational
Sponsor: North-West University, South Africa (Other)
Responsible Party: Principal Investigator, Cristian Ricci, Dr, North-West University, South Africa
Other Study IDs: XXXX1
Record Dates: First submitted 2017-07-06; First posted 2017-07-18 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Diet Modification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: fat intake — Observational study on fat intake and mortality

SUMMARY:
Background Cancer and cardiovascular diseases combined account for more than 50% of the overall mortality burden in the USA. Accumulating evidence indicates that saturated fat intake is related to an increase, while unsaturated fat intake is related to a decrease in all-causes mortality. Thus, current US dietary guidelines recommend a shift from saturated to unsaturated fat.

Objective The aim of the present study was to estimate the mortality risk reduction related to a dietary change from saturated fat to an equal amount of mono or polyunsaturated fat intake.

Design The American National health and nutrition examination surveys conducted between 1999 and 2010 were linked to the 2011 national US death registry resulting in an observational prospective mortality study. Proportional hazards Cox models were used to evaluate the association between saturated, mono-unsaturated and poly-unsaturated fat with all-cause, and cause specific mortality. Substitution analysis was conducted to estimate an iso-caloric substitution of 10% of the energy from dietary fat intake applied to the substitution of saturated fat with an equal amount of energy from mono-unsaturated or poly-unsaturated fat.

ELIGIBILITY:
Inclusion Criteria:

* Included NHANES 1999-2010
* age >= 30 years old

Exclusion Criteria:

* Record not reported in the mortality linked file
* Cancer, type-II diabetes, cardiovascular disease at baseline
* Missing data on covariates used in the model

Ages: 30 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Apparently healthy US adults age>=30
Sampling Method: Probability Sample
Enrollment: 18372 (Actual)
Dates: Start 1999-01-01 (Actual); Primary Completion 2011-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
all causes and specific cause mortality | up to 9 years of observatinal time
  specific cause mortality = cancer and cardiovascular disease

IPD SHARING:
Plan to Share IPD: Yes